CLINICAL TRIAL: NCT03966807
Title: Beyond the Lung Cancer Diagnosis: Leveraging the Oncology Clinic Setting as a Potential Teachable Moment for Actively Smoking Family Members
Brief Title: Beyond the Lung Cancer Diagnosis: Leveraging the Oncology Clinic Setting for Actively Smoking Family Members
Status: Terminated | Type: Observational
Why Stopped: Per institutional and PI recommendation
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Shadia Jalal, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: IUSCC-0670
Record Dates: First submitted 2019-03-18; First posted 2019-05-29 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: lung cancer; caregiver
MeSH Terms: conditions — Lung Neoplasms | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digital-based support: Digital support will consist of referral for the participant to visit https://smokefree.gov, a website which offers a menu of internet- and text-based support options.
  Interventions: Behavioral: Digital-based support
- traditional-based support +nicotine replacement therapy(NRT): Traditional support will consist of participant referral to the Indiana Tobacco Quitline (1-800-QUIT-NOW) which is a telephone hotline that connects participants to Indiana smoking cessation resources.
  Interventions: Behavioral: Traditional-based support + Nicotine replacement therapy (NRT)

INTERVENTIONS:
Behavioral: Digital-based support — Digital support will consist of referral for the participant to visit https://smokefree.gov, a website which offers a menu of internet- and text-based support options.
  Groups: Digital-based support
Behavioral: Traditional-based support + Nicotine replacement therapy (NRT) — Traditional support will consist of participant referral to the Indiana Tobacco Quitline (1-800-QUIT-NOW) which is a telephone hotline that connects participants to Indiana smoking cessation resources.
  Groups: traditional-based support +nicotine replacement therapy(NRT)

SUMMARY:
The purpose of this pilot study is to examine, in an innovative setting, the potential for a lung cancer diagnosis in a loved one to represent a teachable moment for smoking cessation in family members or caregivers who are current smokers. The researchers will identify the willingness and preferred modality for smoking cessation among family members/caregivers in this setting. The researchers will estimate abstinence rates at 4, 8, 12, and 24 weeks..

ELIGIBILITY:
Patient Inclusion Criteria:

1. patient with newly diagnosed lung cancer within the last 6 months of initial diagnosis/confirmation of diagnosis at the study sites
2. Able to provide informed consent
3. Able to speak and read English

Family Member/Caregiver Participant Criteria:

1. Family member or caregiver (defined as first degree relative [parent, sibling, child] or person living in the same household)
2. Family member or caregiver must be a current, active smoker (defined as 10 cigarettes per day for 6 consecutive months).
3. At least 18 years of age at time of study consent
4. Able to provide informed consent
5. Able to speak and read English

Exclusion Criteria:

1. Currently receiving formal tobacco dependence treatment- Nicotine replacement of any kind, varenicycline or Bupropion.
2. Medical condition that precludes proposed pharmacotherapy for smoking cessation : Recent (≤ 2 weeks) myocardial infarction , history of underlying arrhythmias , history of serious or worsening angina pectoris, pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed lung cancers will be identified from the daily patient lists at the thoracic oncology clinics at IUSCC, Roudebush VAMC, and Eskenazi. The study coordinator will screen for newly diagnosed lung cancer patients to identify potential family member/caregiver study participants.
  Patients will be approached and asked whether they have any family members/caregivers who smoke, and if they would be willing to allow the study team to contact those people (or person) with information about the study. For patients who agree and have family members/caregivers present at the clinic visit that day, the study coordinator (or other designated member of the study team) will discuss the purpose of the study and utilize the 5A strategy (Ask, Advice, Assess willingness to quit, Assist, Arrange follow-up) to ascertain interest in participation.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence of self -reported smoking cessation | 4 weeks
7-day point prevalence of self -reported smoking cessation | 8 weeks
7-day point prevalence of self -reported smoking cessation | 12 weeks
7-day point prevalence of self -reported smoking cessation | 24 weeks
Willingness to quit | 4 weeks
Willingness to quit | 8 weeks
Willingness to quit | 12 weeks
Willingness to quit | 24 weeks
Preference for type of cessation intervention modality | 4 weeks
  digital versus traditional support with nicotine replacement therapy [NRT]
Preference for type of cessation intervention modality | 8 weeks
  digital versus traditional support with nicotine replacement therapy [NRT]
Preference for type of cessation intervention modality | 12 weeks
  digital versus traditional support with nicotine replacement therapy [NRT]
Preference for type of cessation intervention modality | 24 weeks
  digital versus traditional support with nicotine replacement therapy [NRT]

SECONDARY OUTCOMES:
Mean change in readiness to quit | Baseline
  Measured via the Readiness to Quit Ladder
Mean change in readiness to quit | 4 weeks
  Measured via the Readiness to Quit Ladder
Mean change in readiness to quit | 8 weeks
  Measured via the Readiness to Quit Ladder
Mean change in readiness to quit | 12 weeks
  Measured via the Readiness to Quit Ladder
Mean change in readiness to quit | 24 weeks
  Measured via the Readiness to Quit Ladder
Mean change in nicotine dependence | Baseline
  Measured via the Heaviness of Smoking Index
Mean change in nicotine dependence | 4 weeks
  Measured via the Heaviness of Smoking Index
Mean change in nicotine dependence | 8 weeks
  Measured via the Heaviness of Smoking Index
Mean change in nicotine dependence | 12 weeks
  Measured via the Heaviness of Smoking Index
Mean change in nicotine dependence | 24 weeks
  Measured via the Heaviness of Smoking Index
Mean change in cigarette use | Baseline
  Measured by by the self-reported number of cigarettes smoked per day
Mean change in cigarette use | 4 weeks
  Measured by by the self-reported number of cigarettes smoked per day
Mean change in cigarette use | 8 weeks
  Measured by by the self-reported number of cigarettes smoked per day
Mean change in cigarette use | 12 weeks
  Measured by by the self-reported number of cigarettes smoked per day
Mean change in cigarette use | 24 weeks
  Measured by by the self-reported number of cigarettes smoked per day

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States